CLINICAL TRIAL: NCT07070635
Title: The Effect of the Fermented Seaweed Enriched Abertay Tea on Vascular Function and Markers of Cardiovascular Risk During Menopause
Brief Title: Abertay Tea for Cardiovascular Health During Menopause
Acronym: AberTeaM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abertay University (Other)
Collaborators: Oshun Labs Ltd (Unknown); UK Research and Innovation (Other)
Responsible Party: Principal Investigator, Sarah Cottin, Lecturer in Nutritional Sciences, Abertay University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EMS9960
Record Dates: First submitted 2025-06-11; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Risk Factor; Vascular Function
Keywords: seaweed; fermented; menopause; vascular function; cardiovascular risk; continuous non invasive arterial pressure

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fermented Seaweed Enriched English Breakfast Tea (Experimental): Nutritional intervention with English Breakfast Tea enriched with Fermented Seaweed
  Interventions: Other: Nutritional intervention with Fermented Seaweed Enriched English Breakfast Tea
- Control Tea (Placebo Comparator): Nutritional intervention with English Breakfast Tea only
  Interventions: Other: Nutritional intervention with Control English Breakfast Tea

INTERVENTIONS:
Other: Nutritional intervention with Fermented Seaweed Enriched English Breakfast Tea — Participants will consume 3 cups of tea per day - spread out during the day, for 8 weeks. For each cup, they will be asked to briefly stir one tea bag (3g tea + 1 g fermented seaweed) into 250mL boiling water and let it brew for 3minutes, before removing the tea bag without squeezing it.
  Arms: Fermented Seaweed Enriched English Breakfast Tea
Other: Nutritional intervention with Control English Breakfast Tea — Participants will consume 3 cups of tea per day - spread out during the day, for 8 weeks. For each cup, they will be asked to briefly stir one tea bag (3g tea) into 250mL boiling water and let it brew for 3minutes, before removing the tea bag without squeezing it.
  Arms: Control Tea

SUMMARY:
The regular consumption of seaweed, as observed in Japan, is associated to a reduced cardiovascular risk and prolonged life expectancy. Interventional studies have shown that brown seaweed consumption can reduce blood pressure, improve glycaemic control and lipoprotein profiles, although this varies with population, dose, duration and the type of seaweed. Brown seaweed appears the most promising to improve cardiovascular risk, due to the presence of specific antioxidants (polyphenols called phlorotannins), pigments (fucoxanthin) and fibre (alginate, fucoidan).

Women see their cardiovascular risk greatly increased when they reach menopause, and seaweed consumption may provide benefits for this population. In the UK, 98% of UK residents drink tea daily (Source UKTIA), with English breakfast tea being the most popular. Providing a tea enriched with beneficial compounds has the potential to improve cardiovascular health in a wide range of the population, including postmenopausal women. Abertay university (Dundee, UK) has recently developed an English Breakfast tea enriched with fermented seaweed, which was found to taste like English breakfast tea. We hypothesise that the consumption of 3 cups a day of the Abertay-developed Tea (AberTea) for 8 weeks, with each tea bag containing 1g of fermented seaweed, will improve vascular function and cardiovascular risk factors in postmenopausal women.

DETAILED DESCRIPTION:
A parallel double-blind randomised controlled trial will be run to test the effects of the AberTea (enriched with fermented seaweed) compared to a control tea on blood pressure and vascular function (primary outcomes) as well as lipoprotein profiles and glycaemic control (secondary outcomes).

Participants will be recruited through internal email circulars, posters and social media amongst Abertay students and staff, and the local community. Volunteers expressing interest will initially be sent an information sheet and a summary of the study by e-mail, with an eligibility questionnaire to fill-in. Volunteers who are eligible will then be invited to attend a short screening session (~20min) during which anthropometric measurements and fasting glucose measurements will be taken, physical activity levels, and important cofactor when examining vascular function, will be assessed using RPAQ. Volunteers who meet the inclusion criteria and sign the consent form will be enrolled in the study and will be randomly allocated to consume 3 cups of Control Tea or AberTea for 8 weeks, they will be asked to not change any other habits, including dietary and physical activity habits.

Participants will then be asked to come back to Abertay fasting for baseline (wk 0) and endpoint (wk 8) measurements. Briefly, vascular and anthropometric measurements will be performed, fasting blood samples will be taken to measure markers of cardiovascular risk, and postmenopausal symptoms will also be assessed.

On visit 1 the participants will be provided with the totality of tea bags needed for the trial (168 tea bags) plus 12 extras, i.e.180 tea bags in total. Regular calls and emails (every 2 weeks) will be maintained between the researchers and participant to ensure compliance. Compliance will be assessed via a tea log sheet provided at the start of intervention, as well as counting the tea bags leftover.

Data will be analysed by analysis of covariance (ANCOVA) of the changes from baseline values, adjusted for ethnicity, age and physical activity levels. Normality of the residuals will be checked for analysis and log transformation of the data will be attempted when required. If the residuals of the log-transformed data are still not normally distributed, non-parametrical analysis will be performed (Mann-Whitney, Kruskal-Wallis). Results will be expressed as means (SD) and changes from baseline as differences between the means with 95% confidence intervals. When data are log transformed, the results will be expressed as geometric means (SD) and the changes as ratios of the geometric means with 95% confidence intervals. All statistical analysis will be carried out with SPSS for Windows (version 29.0, SPSS, Chicago, IL) on the intention-to-treat basis.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal status: no menstrual period over the last 12 months
* Regular tea drinkers (at least once a week), willingness to consume 3 cups of English breakfast tea per day for 8 weeks
* BMI between 18.5 and 39.99 kg/m2

Exclusion Criteria:

* Reported history of CVD (myocardial infarction, angina, venous thrombosis, stroke, dyslipidemia), diabetes (or fasting glucose ≥ 6.1 mmol/L), kidney, liver or bowel disease.
* Recent history of cancer (<1y)
* History indicative of a congenital or acquired platelet or haemostatic defect.
* Presence of gastrointestinal disorder or use of drug, which is likely to alter gastrointestinal motility or nutrient absorption.
* Recent use of hypolipidaemic, antiplatelet or antithrombotic medications
* Impairment of thyroid function
* Current smokers or vapers
* Current self-reported weekly alcohol intake exceeding 14 units
* Current or recent use of hormone replacement therapy (<3 months)
* Recent participation in another clinical trial (<3 months)
* Allergy or intolerance to crustaceans or iodine

Ages: 45 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Continuous Non Invasive Arterial Blood Pressure (CNAP) measurements = Continuous Systolic Blood Pressure | Change from baseline at week 8
  All the non-invasive vascular measurements will be performed in the seated position on the non-dominant arm. The participant will be given a minimum of 5 min rest, time during which a continuous non invasive arterial pressure (CNAP®) monitor will be fitted on their arm and fingers as per the manufacturer's instructions. The participant will be asked to remain as relaxed and calm as possible, so their left arm remains still during the measurements.
  After 5 min rest, a brachial calibration will be performed, followed by the concomitant measurements of CNAP (continuous non-invasive systolic arterial pressure)

SECONDARY OUTCOMES:
Continuous Non Invasive Arterial Blood Pressure (CNAP) measurements = Diastolic Blood Pressure, Mean Arterial Pressure and Pulse; and haemodynamic parameters | Change form baseline to 8 weeks
  All the non-invasive vascular measurements will be performed in the seated position on the non-dominant arm. The participant will be given a minimum of 5 min rest, time during which a continuous non invasive arterial pressure (CNAP®) monitor will be fitted on their arm and fingers as per the manufacturer's instructions. The participant will be asked to remain as relaxed and calm as possible, so their left arm remains still during the measurements. After 5 min rest, a brachial calibration will be performed, followed by the concomitant measurements of CNAP (continuous non-invasive arterial pressure, diastolic, mean), pulse rate, continuous non-invasive cardiac output (CO), stroke volume (SV), and systemic vascular resistance (SVR) for 15min.
Pulse Wave Analysis | Change from baseline at week 8
  The high sampling rate of the CNAP (100Hz) allows the detailed analysis of the pulse waves, providing indices such as the increase in amplitude caused by contraction of the myocardium (AP1), and the return of the reflected wave (AP2), the length of time required for the pulse wave to reach peak systolic pressure (TP1), peak dicrotic pressure (TP2), and the total duration of the cardiac cycle (TPT)
Lipoprotein levels | Change from baseline at week 8
  Serum Total Cholesterol, LDL and HDL will be measured by colorimetric assay
Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) | Change from baseline at week 8
  Based on fasting plasma Insulin and Glucose measurements, using the following formula: [Fasting Insulin (μg/ml)]*[Fasting Glucose (mmol/l)]/22.5

CONTACTS AND LOCATIONS:
Overall Officials: Sarah C Cottin, PhD, Principal Investigator — Abertay University
Locations (1):
- Abertay University, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes